CLINICAL TRIAL: NCT02017067
Title: The Effect of Exercise Training in the Community-dwelling Adults With Chronic Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: FEMH-IRB-101020-E
Record Dates: First submitted 2013-12-05; First posted 2013-12-20 (Estimated); Last update posted 2013-12-20 (Estimated); Status verified 2013-12

CONDITIONS: Osteoporosis; Osteoarthritis
Keywords: Resistance training; musculoskeletal conditions; RFD
MeSH Terms: conditions — Osteoporosis; Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control (No Intervention): Maintain regular physical activity as usual, and received health education material about their disease, importance of nutrition and risks factors.
- hydraulic resistance circuit training (Experimental): 12 weeks resistance training
  Interventions: Procedure: hydraulic resistance circuit training

INTERVENTIONS:
Procedure: hydraulic resistance circuit training — 12 weeks (3 times per week, 40 min circuit) of hydraulic resistance circuit training that consisted of 7 types of equipments for different part of strength training.
  Arms: hydraulic resistance circuit training

SUMMARY:
Previous studies have demonstrated that resistance training (RT) is beneficial to increase muscle strength, improve functional ability and the ability to rapidly produce force, known as the contractile rate of force development (RFD) in older adults. However, much less research has focused on the effect of RT on the lower extremity muscle strength, contractile RFD and impulse in middle-aged and older people with musculoskeletal conditions, especially for osteoporosis (OP) (or osteopenia) or knee osteoarthritis (KOA). Therefore, the purpose of this study was to investigate the effect of RT on the lower extremity muscle strength, RFD and impulse in middle-aged and older people with musculoskeletal conditions, especially for OP and knee OA (KOA). The investigators hypothesized that such a training program would lead to induce not only specific muscle strength enhancement but also an increment in contractile RFD and impulse.

DETAILED DESCRIPTION:
Osteoporosis (OP) and osteoarthritis (OA) are the two most common musculoskeletal conditions in older adults, causing high healthcare costs and negative effects on quality of life. Previous studies have reported that OP and OA has a strong association with sarcopenia, a term defined as age-related involuntary loss of skeletal muscle mass and strength or function.A decline of muscle mass and strength in older adults may limit a variety of activities of daily living (ADLs) and increase morbidity and mortality. However, many ADLs often involve faster limb movements with contraction times of 50 - 200 ms (i.e. sit-to-stand performance and avoiding falls). Therefore, in addition to muscle mass and strength, the ability to rapidly produce force, known as the contractile rate of force development (RFD), and the area under the force-time curve, defined as contractile impulse, seem to be important to adequately characterize the performance of ADLs in older adults. Typically, resistance training (RT) is often prescribed to increase muscle strength, improve functional ability and eliminate much of age-associated muscle atrophy and weakness in a healthy population. Other studies have also shown that implementation of RT can help improve RFD in healthy young and elderly individuals following RT. However, it still unclear that the effect of RT on contractile RFD and impulse in middle-aged and older people with musculoskeletal conditions. Therefore, the aim of this study was to examine the effects on the lower extremity muscle strength, contractile rate of force development (RFD), impulse in middle-aged and older people with osteoporosis (OP)(or osteopenia) or knee osteoarthritis (KOA) after 12 weeks of resistance training.

ELIGIBILITY:
Inclusion Criteria:

(1) 45 years old or older; (2) diagnosed by a physician with osteoporosis (or osteopenia) or/and osteoarthritis; (3) able to participate safely in a moderately vigorous program of physical activity; (4) not previously taken part in any type of resistance training but were all physically capable of entering exercise.

Exclusion Criteria:

(1) a acute or terminal illness, myocardial infarction within 6 months (or other symptomatic coronary artery disease); (2) uncontrolled hypertension (> 150/90 mmHg); (3) fracture in the previous 6 months; (3) diseases or medication affecting neuromuscular function; (4) physical limitation in sports and were advised not to exercise by doctors.

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2012-04; Primary Completion 2013-07 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Maximum voluntary contraction (MVC) | three months
  Muscle strength was measured as maximum voluntary contraction (MVC) of the quadriceps exerted on an isokinetic dynamometer.

SECONDARY OUTCOMES:
Contractile rate of force development (RFD) | three months
  Contractile rate of force development (RFD) was derived as the average slope of the initial phase of the torque-time curve (change in torque/change in time) at 0-30, 50, 100, and 200 ms relative to the onset of contraction.
Impulse | three months
  Contractile impulse was determined as the area under the torque -time curve in the same time intervals of 0-30, 0-50, 0-100, and 0-200 ms relative to the onset of contraction.

CONTACTS AND LOCATIONS:
Overall Officials: Tsung-Ching Lin, Master, Study Chair — Far Eastern Memorial Hospital
Locations (1):
- Tsung-Ching Lin, New Taipei City, Taiwan, Taiwan